CLINICAL TRIAL: NCT06654050
Title: Phase II Study of Alrizomadlin (APG-115) in Subjects With BAP1 Cancer Syndrome and Early-Stage Mesothelioma
Brief Title: Alrizomadlin (APG-115) in Subjects With BAP1 Cancer Syndrome and Early-Stage Mesothelioma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001605; 001605-C
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-08-14

CONDITIONS: Mesothelioma; Malignant Mesothelioma (MM); Early-stage Mesothelioma; Subclinical Mesothelioma; BRCA1-Associated Protein-1 (BAP1) Mutations; Early-stage BAP1-associated Malignancies
Keywords: BRCA1-Associated Protein-1 (BAP1); BAP1 Cancer Syndrome (BCS); BAP1 Cancer Predisposition Syndrome (CPDS); ring finger domains 1 (UHRF1); mdm2 inhibitors (MDM2 inhibitors); p53; DNA methyltransferases 1 (DNMT1); peripheral immune subsets
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/ Arm 1 (Experimental): APG-115
  Interventions: Drug: alrizomadlin

INTERVENTIONS:
Drug: alrizomadlin — Alrizomadlin (APG-115) oral tablets (150 mg) taken every other day on Days 1, 3, 5, 7, 9, 11, and 13 of every cycle (1 cycle=21 days) for 8 cycles (i.e., Course 1). Individuals with stable or responding disease may receive an additional 8 cycles (i.e., Course 2). Maximum (total) of 2 treatment courses.

SUMMARY:
Background:

Mesothelioma is a rare cancer typically caused by exposure to asbestos and related fibers. Most people with mesothelioma survive less than 5 years after diagnosis. About 3000 people in the United States die from this disease each year. People with inherited mutations in the BAP1 gene [called BAP1 Cancer Syndrome (BCS)] are more likely to develop mesothelioma and other cancers such as melanomas and renal cell carcinomas without asbestos exposure. Almost all people with BCS develop multiple cancers, of which mesothelioma is the most commonly observed.

Objective:

To test a study drug (APG-115) in participants with BAP1 Cancer Syndrome (BCS) and early-stage mesothelioma.

Eligibility:

People aged 18 years and older with germline BAP1 mutations and early-stage mesothelioma that does not yet need standard treatment are eligible for protocol enrollment. Participants will be required to also enroll in NIH protocols 20-C-0106 and 06-C-0014 which allow for pre- and post-treatment biopsies and bloodwork to be obtained for additional research studies.

Design:

Participants will be screened. They will have a physical exam with blood tests. Their medical records will be reviewed. They will have imaging scans and tests of their heart and lung functions. A procedure using a flexible tube with a camera and light will be inserted into the participant s chest and abdomen through a small cut to look at the tumors and to collect a tissue sample (biopsy).

APG-115 capsules are taken by mouth. Participants will take the drug at home every other day for the first 13 days of the 21-day treatment cycles.

On the first day of each cycle, researchers will call or email participants to check on their health.

Participants will have blood tests 2 times a week during the first 2 cycles; after that, the blood tests will be weekly. These blood tests can be done at a local medical facility or at the NIH Clinical Center.

Participants may continue treatment for up to 16 cycles.

Imaging scans, biopsy, and other tests will be repeated after 8 and 16 cycles.

DETAILED DESCRIPTION:
Background:

* Mutations involving BRCA1-Associated Protein-1 (BAP1), a nuclear deubiquitinase involved in epigenetic regulation of gene expression, DNA repair, and cellular energetics, have emerged as one of the most common somatic mutations in malignant mesotheliomas.
* Germline mutations involving BAP1 predispose individuals to mesotheliomas and a variety of other malignancies including melanomas, as well as lung, renal, gastric, breast, and hepatobiliary carcinomas.
* The cancer penetrance of germline BAP1 mutations is nearly 100%, and most patients develop multiple synchronous or metachronous neoplasms.
* Mesotheliomas are the most common malignancies diagnosed in subjects with BAP1 Cancer Syndrome (BCS), previously known as BAP1 Cancer Predisposition Syndrome (CPDS).
* Although clinically evident mesotheliomas arising in the context of germline BAP1 mutations tend to be more indolent than more common, sporadic mesotheliomas, the natural history of early-stage mesotheliomas in subjects with BAP1 BCS is unknown.
* Presently there are no established guidelines for the treatment of subclinical malignancies in subjects with BAP1 BCS.
* Ubiquitin-like with plant homeodomain and ring finger domains 1 (UHRF1) is a master regulator of DNA methylation and genome integrity in normal cells.
* Up-regulation of UHRF1 during malignant transformation induces widespread epigenomic perturbations including global DNA hypomethylation and paradoxical site-specific DNA hypermethylation of tumor suppressor genes.
* Dysregulation of DNA methylation induces genomic instability and enhances growth as well as invasion and metastatic potential of cancer cells and promotes an immunosuppressive tumor micro-environment (TME).
* Up-regulation of UHRF1 is an early event during mesothelioma development, and UHRF1 over-expression is associated with markedly decreased survival in mesothelioma patients.
* Biochemical inhibition of UHRF1 expression inhibits the growth of mesothelioma cells invitro and in-vivo.
* UHRF1 expression can be repressed by mdm2 inhibitors which activate p53 signaling. In addition to direct effects on cancer cells, mdm2 inhibitors can reprogram TMEs thereby promoting more effective antitumor immune responses.
* APG-115 is an oral, highly potent, mdm2 inhibitor that is in clinical development.
* Conceivably APG-115 therapy can arrest or delay the progression of subclinical/early stage mesotheliomas in subjects with BAP1 BCS.

Objective:

-To determine stabilization or disease improvement rates in participants with early-stage mesotheliomas arising in the context of BAP1 Cancer Syndrome (BCS) following APG-115 treatment

Eligibility:

* History of germline BRCA1-Associated Protein-1 (BAP1) mutations.
* Histologically confirmed subclinical/early-stage mesotheliomas.
* The extent of the disease must be insufficient to warrant approved front-line standard-of care therapies (surgery, chemotherapy, immunotherapy).
* Age >= 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status <=1.
* Willingness to undergo pre- and post-treatment, minimally invasive thoracoscopy, and/or laparoscopy to assess treatment response.
* Adequate cardiac, renal, hepatic, and hematopoietic function.

Design:

* Participants with subclinical, early-stage mesotheliomas will undergo baseline imaging studies followed by minimally invasive thoracoscopy and/or laparoscopy to document the extent of the disease and obtain biopsies for pharmacodynamic (PD) endpoints.
* Participants will start oral APG-115 at a fixed dose and schedule (150 mg on Days 1, 3, 5,7, 9, 11, and 13 of a 21-day cycle) and will continue this regimen for 8 cycles.
* After eight cycles, participants will undergo repeat imaging and minimally invasive thoracoscopy and/or laparoscopy to determine treatment response and obtain tissue for response endpoints.
* Participants with stable disease or disease regression will be offered an additional 8 cycles of APG-115 treatment.
* Approximately 13 participants will be administered investigational therapy on this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:
* History of germline BRCA1-Associated Protein-1 (BAP1) mutations.
* Histologically confirmed by NCI Laboratory of Pathology (LP) subclinical/early-stage mesotheliomas.
* Participants with other early-stage BAP1-associated malignancies in addition to subclinical, early-stage mesotheliomas are eligible for the study.
* The extent of the disease (Tx by clinical staging criteria) must be insufficient to warrant approved front-line standard of care (SOC) therapies (surgery, chemotherapy, immunotherapy). Participants with clinical T1 tumors are eligible for protocol if they have been offered and have refused front-line SOC therapy.
* Age >=18 years.
* Evaluable disease as confirmed by minimally invasive (videoscopic) assessment (thoracoscopy and/or laparoscopy with biopsy).
* Willingness to undergo pre- and post-treatment minimally invasive thoracoscopy and/orlaparoscopy to assess treatment response.
* Willingness to co-enroll on 20-C-0106 (Prospective Evaluation of High Resolution Dual Energy Computed Tomographic Imaging, Noninvasive (Liquid) Biopsies, and Minimally Invasive Surgical Surveillance for Early Detection of Mesotheliomas in Patients with BAP1 Tumor Predisposition Syndrome) and 06-C-0014 (Prospective Evaluation of Genetic and Epigenetic Alterations in Patients with Thoracic) to enable collection/processing of tumor, blood and normal pleura).
* ECOG performance status <=1
* Adequate pulmonary reserve evidenced by forced expiratory volume (FEV)1 and diffusing capacity of the lungs for carbon monoxide (DLCO) >=35% predicted on screening pulmonary function testing (PFTs).
* Oxygen saturation >=92% on room air by pulse oximetry at screening.
* Adequate renal, hepatic, and hematopoietic function as defined below:

  * leukocytes >= 3,000/micro L
  * absolute neutrophil count >=1,500/micro L (without transfusion or cytokine support within 2 months prior to study treatment initiation)
  * absolute lymphocyte count > 800/micro L
  * platelets >= 100,000/micro L and < 1,200,000/micro L
  * prothrombin time (PT) no more than 2 seconds above the upper limit of normal (ULN)
  * total bilirubin < 1.5 X institutional ULN OR direct bilirubin <= 1 ULN for participants with total bilirubin >= 1.5 ULN serum albumin >=2.0 mg/dL
  * aspartate aminotransferase (AST) <=2.5 X institutional ULN
  * alanine aminotransferase (ALT) <= 2.5 X institutional ULN
  * estimated glomerular filtration rate (eGFR) >=60 mL/min/1.73 m2.
* Individuals of child-bearing potential (IOCBP) and those able to father a child must agree to use an effective method of contraception (barrier, hormonal, intrauterine device (IUD), surgical sterilization) from the study entry and up to 3 months after the last dose of APG-115.
* Nursing (i.e., breastfeeding/chest feeding) participants must be willing to discontinue nursing from study treatment initiation through 4 weeks after the last dose of the study drug.
* The ability of a participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants with any cancers requiring front-line standard of care treatment.
* Clinically significant cardiovascular/cerebrovascular disease as follows: cerebral vascular accident/stroke within 6 months prior to study treatment initiation, myocardial infarction within 6 months prior to study treatment initiation unless revascularized post infarction and cleared by cardiology consultants.
* Unstable angina, congestive heart failure (New York Heart Association Classification Class >= II (https://manual.jointcommission.org/releases/TJC2016A/DataElem0439.html#:~:text=Class%20II%20%2D%20Mild%20symptoms%20(mild,Class%20IV%20%2D%20Severe%20limitations.), serious cardiac arrhythmia, clinically significant bleeding or clinically significant pulmonary embolism at screening.
* QTcF interval > than the 470 ms.
* Therapeutic anticoagulation within 2 weeks prior to study treatment initiation. Note: Oral agents and Lovenox, etc., are monitored by factor 10 levels, not PT or partial thromboplastin time (PTT).
* Participants receiving inhibitors or inducers of CYP3A4/3A5 as well as participants receiving P-glycoprotein inhibitors within 2 weeks prior to study treatment initiation treatment initiation

(https://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/ucm093664.htm#table2-2,table3-3,table5-2,

* Positive Hepatitis A (HAV) serological test, positive Hepatitis B (HBV) serological test, or positive Hepatitis C (HCV) serological test with detected quantitative HCV RNA at screening.
* Participants seropositive for human immunodeficiency virus (HIV) infection.
* Active infections requiring systemic therapy.
* Immunosuppressive medications within 4 weeks prior to study treatment initiation except non-systemic corticosteroids.
* Positive beta human chorionic gonadotropin (beta-HCG) serum or urine pregnancy test performed in individuals of childbearing potential at screening.
* Uncontrolled intercurrent illness evaluated by medical history and physical exam or situation that is not stable (e.g., recent hospitalization, Emergency Room visit or undergoing medication changes) that would potentially increase in risk of participant.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine stabilization or disease improvement rates in participants with early-stage mesotheliomas arising in the context of BAP1 Cancer Syndrome (BCS) following APG-115 treatment | baseline, and after every 8 treatment cycles (Course 1 and Course 2)
  Fraction of evaluable participants who are able to have stabilization or improvement of disease will be reported along with a 95% confidence interval. Response rates will be calculated as the percent of participants whose best response is a stabilization or improvement of disease.

SECONDARY OUTCOMES:
To evaluate the safety of APG-115 | starts at initiation of study drug, assessed Days 1 of every cycle, and through 30 days (safety visit) after the last study drug administration
  Safety and tolerability of the agents will be evaluated by reviewing the AEs and reporting events as required. Toxicity information recorded will include the type, severity, time of onset, time of resolution, and probable association with the study regimen.

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded will be shared upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers within 10 years after the completion of the primary endpoint by contacting the Principal Investigator.
Access Criteria: Data from this study may be requested by contacting the PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001605-C.html